CLINICAL TRIAL: NCT04501159
Title: Observational Study to Assess pH and Hypoxia During Haemodialysis
Brief Title: pH, Hypoxia and Haemodialysis
Acronym: pHHd
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Coventry University (Other)
Collaborators: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Principal Investigator, Scott McGuire, Post-Doctoral Researcher, Coventry University
Other Study IDs: 281803
Record Dates: First submitted 2020-07-29; First posted 2020-08-06 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: ESRD: End-stage renal disease; ABG: Arterial blood gases; NICOM: Non-invasive cardiac output monitour; HD: Haemodialysis; WBC: white blood cell
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- End-stage renal disease (ESRD): Patients with end-stage renal disease undergoing regular haemodialysis 3 times weekly.The investigation will measure cardiac output (CO), oxygen saturation (SaO2), arterial blood gases (ABG) and white blood cell (WBC) count during HD to assess changes in haemodynamics, pH, leukostasis and hypoxia. Patients undergoing regular HD will be recruited with arterial blood samples for gas analysis drawn over three consecutive HD treatments. Arterial samples will be taken at the start, 15 minutes and end of HD treatment for ABG and WBC analysis. Dialysis membrane, ultrafiltration volume, serum and dialysate bicarbonate levels will also be recorded. Regression analysis will be performed with pH, ABG and SaO2. A subset of patients will be used to assess an if cardiac output, WBC or pH better predicts PaO2 during HD.
  Interventions: Other: blood sample pre, during and post HD; Device: Non invasive cardiac output assessment

INTERVENTIONS:
Other: blood sample pre, during and post HD — Assessment of ABG pre, during and post HD
Device: Non invasive cardiac output assessment — Four ECG style electrodes are placed on the thorax which indirectly measures cardiac output.
  Other Names: NICOM

SUMMARY:
End-stage renal disease typically requires haemodialysis to help replace kidney function. However, changes in oxygen uptake during haemodialysis have been linked to increased all-cause mortality. This complication of haemodialysis is linked to decreasing fluid volume, compromising blood flow to tissue and leukostasis within pulmonary tissue. However, an alternative cause of reduced oxygen availability (hypoxia) during haemodialysis is acute alkalosis. Alkalosis during haemodialysis can cause hypoxia via dysregulated ventilation and impaired ability for tissue to extract oxygen. Despite strong rationale for these mechanisms, few studies have fully explored causes of hypoxia during haemodialysis. Greater understanding may help to mitigate the risk associated with this vital treatment option.

The study will comprise of end-stage renal disease patients who regularly undergo haemodialysis. Three blood samples will be attained before, during and after haemodialysis to assess arterial blood gases. In a small subset of patients, white blood cell (WBC) count and cardiac output will be assessed via a non-invasive cardiac output monitor during treatment. Regression analysis will be performed to help identify predictors of hypoxia during haemodialysis. Patient burden is negligible, with blood samples attained from the dialyser as part of routine treatment. In the patients who agree for cardiac output assessment, the patient will be required to have four small noninvasive sensor pads placed on the chest. Patients will be assessed over 3 consecutive treatments during a single week.

DETAILED DESCRIPTION:
Alkalosis may explain multiple complications of HD treatment, most notably hypoxemia. Despite a strong rationale for these mechanisms, current consensus suggests ischaemia as the predominant catalyst for hypoxia with HD. However, few studies have characterised pH changes during HD with many using serum bicarbonate as a proxy of pH status. Nevertheless, these studies predominantly indicate acute alkalosis occurrence with HD. Despite these findings, few HD units individualise their bicarbonate prescription or assess pH prior to treatment. Of 554 dialysis facilities worldwide, 49% did not individualise bicarbonate prescriptions. Non-individualised bicarbonate prescription risks sub-therapeutic serum bicarbonate levels and sub-clinical hypoxemia during HD. Assumption of acidosis and consistent baseline pH prior to each HD session may further risk acute alkalosis with HD. Indeed, a normal pH was identified in 26 ESRD patients on commencing HD whilst prescribed dialysate bicarbonate of 32 mmol/L (7.38 ± 0.06) or 26 mmol/L (7.35 ± 0.06). However, pH increased throughout HD with acute alkalosis within the 32 mmol/L group (7.48 ± 0.05). These data, suggest individualised assessment of pH prior to HD could mitigate alkalosis and subsequent hypoxemia. However, small cohorts, limited studies of pH changes over consecutive HD treatments, and few studies of links between hypoxemia and pH limit current understanding. This study therefore aims to explore pH changes and occurrence of hypoxia with HD.

Adult patients (18+) will be recruited irrespective of age, gender, or ethnicity. Due to the observational nature of the study, no personal benefits will be expressed to the patient. Signed consent will be attained from a patient after a minimum of 24hrs has been provided on receipt of the participation information sheet. Any questions will be clearly answered prior to obtaining consent from the patient. Only patients who have full capacity to give consent and full understanding of the purpose and procedures of the study will be recruited.

There is no foreseen risk to the patient from the study. All blood samples are attained via arterial-venous catheter which is inserted prior to treatment as part of the patient's routine haemodialysis. In the small subset of patients who have their cardiac output assessed, the use of four small non-invasive sensors poses no additional discomfort, risk or restriction throughout routine haemodialysis treatment. In a previous project using the noninvasive cardiac output monitor (NICOM), no patient expressed any discomfort whilst using the device during haemodialysis.

All patients involved in the project will be anonymised with a study number for data collection purposes. No identifiable information will be used during post-hoc analysis. Signed consent forms or any other identifiable data will be securely logged within the study site file and secured within the renal research office. Only the chief investigator and renal research nurses will be aware of patient involvement in the study. Access to identifiable data will be strictly limited to the chief investigator.

There is no conflict of interest from the chief investigator or other members of the research team that may influence the study. After completion of the study, data will be compiled and drafted for scientific publication with all data securely archived within the study site file at the renal research department. Any patient expressing interest in the study findings will be provided with the appropriate information verbally or by a written summary of findings.

All blood samples will consist of ~1.5ml which will be analysed immediately after sampling. Samples will subsequently be disposed of immediately after analysis and not be used for any subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

* On haemodialysis for at least 3 months.
* Haemodialysis 3 times per week.
* Age 18 years or older.

Exclusion Criteria:

* Central venous catheter.
* Planned kidney transplant during the duration of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End-stage renal disease patients will be recruited from the University Hospitals Coventry & Warwickshire hemodialysis unit identified by the research team and renal medical professionals.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-08-21 (Actual); Study Completion 2021-12-29 (Estimated)

PRIMARY OUTCOMES:
To assess change from baseline to end of haemodialysis in pH. | Change in pH pre to post HD over 3 separate HD treatments in a single week.
  Blood samples will be collected in heparinized syringes via HD catheter from end-stage renal disease patients before commencing HD and on HD completion. Arterial blood pH will be determined by ABG analyser immediately after blood sample collection. Patients will be assessed for ABG during a typical week (3 days) of HD treatment.
To assess change from baseline to end of haemodialysis in PaO2. | Change in PaO2 pre to post HD over 3 separate HD treatments in a single week.
  Blood samples will be collected in heparinized syringes via HD catheter from end-stage renal disease patients before commencing HD and on HD completion. Arterial oxygen tension (PaO2) will be determined by ABG analyser immediately after blood sample collection. Patients will be assessed for ABG during a typical week (3 days) of HD treatment.

SECONDARY OUTCOMES:
To assess changes in pH status over a standard three session HD treatment week assessed via ABG. | Before and after HD over 3 separate treatments in a single week.
  To assess the number of patients within an alkalemia state post HD.
To assess if pH is a better predictor of hypoxia during HD than cardiac output. | Assessed before, during (15 mins HD) and after HD on first treatment of the week.
  Cardiac output, leukopenia and pH status have been described to contribute to hypoxia during HD. Regression analysis will determine which, if any, better predicts hypoxia during HD.

CONTACTS AND LOCATIONS:
Overall Officials: Scott McGuire, PhD, Principal Investigator — Coventry University
Locations (2):
- United Kingdom (2):
  - UHCW, Coventry, Warwickshire
  - University Hospital Coventry and Warwickshire, Coventry, West Midlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGuire S, Horton EJ, Renshaw D, Jimenez A, Krishnan N, McGregor G. Hemodynamic Instability during Dialysis: The Potential Role of Intradialytic Exercise. Biomed Res Int. 2018 Feb 27;2018:8276912. doi: 10.1155/2018/8276912. eCollection 2018. PMID 29682559
- [Background] Yap JC, Wang YT, Poh SC. Effect of oxygen on breathing irregularities during haemodialysis in patients with chronic uraemia. Eur Respir J. 1998 Aug;12(2):420-5. doi: 10.1183/09031936.98.12020420. PMID 9727795
- [Background] Assa S, Hummel YM, Voors AA, Kuipers J, Westerhuis R, Groen H, Bakker SJ, Muller Kobold AC, van Oeveren W, Struck J, de Jong PE, Franssen CF. Hemodialysis-induced regional left ventricular systolic dysfunction and inflammation: a cross-sectional study. Am J Kidney Dis. 2014 Aug;64(2):265-73. doi: 10.1053/j.ajkd.2013.11.010. Epub 2013 Dec 21. PMID 24364893
- [Background] Buchanan C, Mohammed A, Cox E, Kohler K, Canaud B, Taal MW, Selby NM, Francis S, McIntyre CW. Intradialytic Cardiac Magnetic Resonance Imaging to Assess Cardiovascular Responses in a Short-Term Trial of Hemodiafiltration and Hemodialysis. J Am Soc Nephrol. 2017 Apr;28(4):1269-1277. doi: 10.1681/ASN.2016060686. Epub 2016 Nov 10. PMID 28122851
- [Background] Dasselaar JJ, Slart RH, Knip M, Pruim J, Tio RA, McIntyre CW, de Jong PE, Franssen CF. Haemodialysis is associated with a pronounced fall in myocardial perfusion. Nephrol Dial Transplant. 2009 Feb;24(2):604-10. doi: 10.1093/ndt/gfn501. Epub 2008 Sep 4. PMID 18775808
- [Background] Kossari N, Hufnagel G, Squara P. Bioreactance: a new tool for cardiac output and thoracic fluid content monitoring during hemodialysis. Hemodial Int. 2009 Oct;13(4):512-7. doi: 10.1111/j.1542-4758.2009.00386.x. Epub 2009 Sep 16. PMID 19758300
- [Background] Misra M. Pro: Higher serum bicarbonate in dialysis patients is protective. Nephrol Dial Transplant. 2016 Aug;31(8):1220-4. doi: 10.1093/ndt/gfw259. Epub 2016 Jul 13. PMID 27411723
- [Background] Tentori F, Karaboyas A, Robinson BM, Morgenstern H, Zhang J, Sen A, Ikizler TA, Rayner H, Fissell RB, Vanholder R, Tomo T, Port FK. Association of dialysate bicarbonate concentration with mortality in the Dialysis Outcomes and Practice Patterns Study (DOPPS). Am J Kidney Dis. 2013 Oct;62(4):738-46. doi: 10.1053/j.ajkd.2013.03.035. Epub 2013 May 24. PMID 23707043
- [Background] Saravanan P, Davidson NC. Risk assessment for sudden cardiac death in dialysis patients. Circ Arrhythm Electrophysiol. 2010 Oct;3(5):553-9. doi: 10.1161/CIRCEP.110.937888. No abstract available. PMID 20959609
- [Background] Gabutti L, Ferrari N, Giudici G, Mombelli G, Marone C. Unexpected haemodynamic instability associated with standard bicarbonate haemodialysis. Nephrol Dial Transplant. 2003 Nov;18(11):2369-76. doi: 10.1093/ndt/gfg383. PMID 14551368